CLINICAL TRIAL: NCT06572735
Title: Study on the Relative Dose Intensity of PARP Inhibitors in Real-life on a Population of Patients Over 70 Years With Advanced Ovarian Cancer
Acronym: PARIB-OLD-PRO²
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0912
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
Keywords: Cancer; ovary; PARP inhibitors; toxicity; elder patients
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Geriatric Assessment; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with advanced ovarian cancer: Patients of 70 years and elder with an advanced ovarian cancer who are scheduled to start a maintenance therapy with PARP inhibitors for the first time. The PARP inhibitors are administrated according to the marketing authorization and will be Olaparib (which may by administrated in combination with Bevacizumab) and Niraparib. There is no specific medical visit for this study, patient are followed in a routine care. Some medical data about the disease follow-up will be collected at inclusion and at each visit, every 3 months over a 12-months period. Furthermore, two quality of life surveys (OV28 and ELD14) and one geriatric assessment will be performed at each visit every 3 months and one 8ml-blood sample will be done at inclusion, and after 6 and 12 months of PARP inhibitors treatment.
  Interventions: Other: QoL surveys; Other: Geriatric assessment (G-CODE); Biological: Blood sampling

INTERVENTIONS:
Other: QoL surveys — 2 quality of life surveys (OV28 and ELD14) will be completed by patients every 3 months during a 12-month period
Other: Geriatric assessment (G-CODE) — A geriatric assessment (G-CODE) will be performed by the research staff every 3 months during a 12-month period
Biological: Blood sampling — A supplementary volume of blood will be collected from a routine blood sample (8 mL) at 3 different time points : one at inclusion, one 6 and 12 months after the beginning of PARP inhibitors treatment. Genetic lab test will be performed to assess whether there is a specific genetic signature for PARP inhibitors toxicity.

SUMMARY:
Poly(ADP-ribose) polymerase (PARP) inhibitors are anti-cancer treatments that induce preferential tumor cell death. Their efficacy has been demonstrated in many tumor models, primarily in advanced ovarian cancer. PARP inhibitors also exhibit a particular toxicity, damaging the hematopoietic tissue. With age, pharmacokinetic changes or a reduction in medullary cavity may increase these toxicities and may lead to dose reductions/postponements or premature discontinuation of PARP inhibitors, which may impact the efficacy of treatment. Close biological monitoring must be carried out to limit these toxicities, in most cases anemia, thrombocytopenia and neutropenia. Until now, the geriatric factors impacting the tolerance and uptake of PARP inhibitors in the elderly patient population with advanced ovarian cancer are not clearly established. It is therefore necessary to have prospective real-life data in order to support patients in a decision-making process on whether or not to continue such treatments.

PARIB-OLD-PRO² will evaluate the association between various clinical, biological, and geriatric factors and the relative dose intensity (RDI) of therapy by PARP inhibitors. This is a prospective, multicenter longitudinal and non-interventional study and will involve a population of 50 patients, aged 70 years and elder, with advanced ovarian cancer who are scheduled to start a therapy with PARP inhibitors for the first time. The aim of the study is to better understand the effects of PARP inhibitors on a elderly population, knowledge of the genetic and clinical determinants of PARP inhibitors toxicity in this specific population and an optimal management of this therapy related adverse events in order to maintain an RDI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Histologically or cytologically confirmed diagnosis of advanced ovarian cancer (FIGO stage III or IV)
* PARP inhibitors -naive patient who need to initiate maintenance treatment with PARP inhibitors for the first time (according the the marketing authorization)
* Patient with a life expectancy of more then 3 months
* Informed patient which does not oppose to participate to the study

Exclusion Criteria:

* Prior treatment with PARP inhibitors
* Patient incapable to take oral tablets/capsules
* Participation in a drug trial that does not authorize concurrent participation in another trials
* Person unable to attend scheduled examinations/appointments as part of routine care for geographical, social or psychological reasons
* Concomitant cancer or f cancer history (other than those included in the inclusion criteria) treated and considered cured for less than 2 years. However, patients with the following pathologies are eligible:

  * Basal cell carcinoma or non-invasive cutaneous squamous cell carcinoma
  * Stage 1B or less cervical carcinoma
  * Non-invasive superficial bladder cancer

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of 70 years and elder with an advanced ovarian cancer who are scheduled to start a maintenance therapy with PARP inhibitors for the first time. The necessary number of patients in the study is 50.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Relative dose intensity of the PARP inhibitors treatment | at 12 months
  Ratio of the delivered PARP inhibitors dose intensity to the planned dose intensity at the beginning of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claire FALANDRY, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (9):
- France (9):
  - Centre Hospitalier Universitaire d'Amiens Picardie Site Sud, Amiens
  - Centre de lutte contre le cancer Jean Perrin, Clermont-Ferrand
  - Groupe Hospitalier Public Sud de l'Oise, Creil
  - Centre Georges François Leclerc, Dijon
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - Service Hôpital de jour / Oncologie Médicale, Hôpital de la Croix Rousse, Lyon
  - Service de Gériatrie, Hôpital Dr Frédéric Dugoujon, Lyon
  - Service Oncologie Médicale, Hôpital Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie et d'Hématologie Universitaire de Saint Etienne, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No